CLINICAL TRIAL: NCT02911753
Title: Feasibility and Acceptability of a Beverage Intervention for Hispanic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1606621176
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Hypercholesterolemia; Hyperglycemia; Hypertriglyceridemia
MeSH Terms: conditions — Obesity; Hypercholesterolemia; Hyperglycemia; Hypertriglyceridemia | interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mediterranean Lemonade Consumption (Experimental): All participants will be asked to consume 32 ounces daily of Mediterranean Lemonade. The beverage will be previously prepared and packaged by study personnel. Participants will receive their beverage supply on a weekly basis for a total of six weeks.
  Interventions: Other: Mediterranean Lemonade
- Green Tea Consumption (Experimental): All participants will be asked to consume 32 ounces daily of Green Tea. The beverage will be previously prepared and packaged by study personnel. Participants will receive their beverage supply on a weekly basis for a total of six weeks.
  Interventions: Other: Green Tea
- Flavored Water Consumption (Placebo Comparator): All participants will be asked to consume 32 ounces daily of Flavored Water. The beverage will be previously prepared and packaged by study personnel. Participants will receive their beverage supply on a weekly basis for a total of six weeks.
  Interventions: Other: Flavored Water

INTERVENTIONS:
Other: Mediterranean Lemonade — All participants will be advised to consume all of the beverage assigned (mediterranean lemonade) on a daily basis (rather than save up and consume large amounts on fewer days). The beverages will be prepared in advance by study personnel, refrigerated, and distributed to study participants on a weekly basis. Participants will be provided a daily 32-ounce beverage container for beverage consumption and instructed to clean the container nightly. Participants will also be asked to keep a log of completion of beverage on a daily basis and instructions regarding intake of other beverages will be provided.
  Other Names: Beverage Consumption Intervention
  Arms: Mediterranean Lemonade Consumption
Other: Green Tea — All participants will be advised to consume all of the beverage assigned (green tea) on a daily basis (rather than save up and consume large amounts on fewer days). The beverages will be prepared in advance by study personnel, refrigerated, and distributed to study participants on a weekly basis. Participants will be provided a daily 32-ounce beverage container for beverage consumption and instructed to clean the container nightly. Participants will also be asked to keep a log of completion of beverage on a daily basis and instructions regarding intake of other beverages will be provided.
  Other Names: Beverage Consumption Intervention
  Arms: Green Tea Consumption
Other: Flavored Water — All participants will be advised to consume all of the beverage assigned (flavored water) on a daily basis (rather than save up and consume large amounts on fewer days). The beverages will be prepared in advance by study personnel, refrigerated, and distributed to study participants on a weekly basis. Participants will be provided a daily 32-ounce beverage container for beverage consumption and instructed to clean the container nightly. Participants will also be asked to keep a log of completion of beverage on a daily basis and instructions regarding intake of other beverages will be provided.
  Other Names: Beverage Consumption Intervention
  Arms: Flavored Water Consumption

SUMMARY:
This study aims to 1) assess the feasibility and acceptability of a prescribed beverage intervention in 50 obese Hispanic adults ages 18-64 years over 6 weeks; and 2) assess preliminary effects of the beverage intervention on cholesterol and triglyceride levels as well as other markers of health such as blood pressure, glucose and markers of inflammation. This project, if successful, will provide early evidence that targeting dietary behavior around beverage intake could be a novel and easily adopted approach to reduce the burden or delay the onset of metabolic abnormalities in obese Hispanic adults. The expected outcome of the proposed project is the identification of feasible and appropriate beverage intervention strategies to improve engagement and adherence to dietary modification approaches for control of metabolic health indicators in this vulnerable ethnic group.

DETAILED DESCRIPTION:
In the U.S., Hispanics have the highest rates of overweight and obesity when compared to other racial/ethnic groups placing them at a greater risk for obesity-related disease. Yet, current literature is limited to information on best practices to engage Hispanics in health-promoting lifestyle interventions. Without this information the health consequences associated with obesity, including high blood pressure, elevated blood glucose and high cholesterol, will continue. Evidence exists to support diet-specific behavioral interventions in reducing obesity-related health risks. Among the more adoptable interventions to date are efforts targeting beverage intake. Yet, there are limited data to suggest these approaches are effective for Hispanics despite this being the fastest growing and highest burdened group for obesity-related disease within the U.S. population.

This study aims to 1) assess the feasibility and acceptability of a prescribed beverage intervention in 50 obese Hispanic adults ages 18-64 years over 6 weeks; 2) assess preliminary effects of the beverage intervention on cholesterol and triglyceride levels as well as other markers of health such as blood pressure, glucose and markers of inflammation. This project, if successful, will provide early evidence that targeting dietary behavior around beverage intake could be a novel and easily adopted approach to reduce the burden or delay the onset of metabolic abnormalities in obese Hispanic adults. The expected outcome of the proposed project is the identification of feasible and appropriate beverage intervention strategies to improve engagement and adherence to dietary modification approaches for control of metabolic health indicators in this vulnerable ethnic group.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic
* 18-64 years of age
* BMI between 30 to 50.0 kg/m²
* Ability to participate in and provide informed consent.
* Speak, read, and write either English and/or Spanish

Exclusion Criteria:

* Diagnosis of diabetes mellitus
* History of liver disease
* Current medication for glucose control, cholesterol control; uncontrolled BP
* Current eating disorders such as anorexia nervosa, bulimia, etc. (likely to make adherence to prescribed beverage intake difficult)
* Current alcohol or substance abuse
* Currently treated for psychological issues (i.e. depression, bipolar disorder, etc.), taking psychotropic medications with the previous 12 months, or hospitalized for depression within the previous 5 years
* Report exercise on ≥3 days per week for ≥ 20 minutes per day over the past 3 months
* Report weight loss of ≥5% or participating in a weight reduction diet program in the past 3 months
* Report plans to relocate to a location that limits their access to the study site or having employment, personal, or travel commitments that prohibit attendance to all of the scheduled assessments
* Report consumption of ≥ 1 cup of green tea daily and not willing to complete 2 week run-in period
* Report consumption of ≥ 1 cup of citrus fruit daily and not willing to complete 2 week run-in period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Garcia, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Collaboratory for Metabolic Disease Prevention and Treatment, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Zheng XX, Xu YL, Li SH, Liu XX, Hui R, Huang XH. Green tea intake lowers fasting serum total and LDL cholesterol in adults: a meta-analysis of 14 randomized controlled trials. Am J Clin Nutr. 2011 Aug;94(2):601-10. doi: 10.3945/ajcn.110.010926. Epub 2011 Jun 29. PMID 21715508
- [Background] Hakim IA, Hartz V, Harris RB, Balentine D, Weisgerber UM, Graver E, Whitacre R, Alberts D. Reproducibility and relative validity of a questionnaire to assess intake of black tea polyphenols in epidemiological studies. Cancer Epidemiol Biomarkers Prev. 2001 Jun;10(6):667-78. PMID 11401918
- [Derived] Garcia DO, Morrill KE, Aceves B, Valdez LA, Rabe BA, Bell ML, Hakim IA, Martinez JA, Thomson CA. Feasibility and acceptability of a beverage intervention for Hispanic adults: results from a pilot randomized controlled trial. Public Health Nutr. 2019 Mar;22(3):542-552. doi: 10.1017/S1368980018003051. Epub 2018 Nov 19. PMID 30451147
- [Derived] Morrill KE, Aceves B, Valdez LA, Thomson CA, Hakim IA, Bell ML, Martinez JA, Garcia DO. Feasibility and acceptability of a beverage intervention for Hispanic adults: a protocol for a pilot randomized controlled trial. Nutr J. 2018 Feb 9;17(1):16. doi: 10.1186/s12937-018-0329-y. PMID 29426328

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mediterranean Lemonade Consumption | Green Tea Consumption | Flavored Water Consumption
Started | 21 | 19 | 10
Completed | 18 | 16 | 10
Not Completed | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Flavored Water: All participants were advised to consume all of the beverage assigned (flavored water) on a daily basis (rather than save up and consume large amounts on fewer days). The beverages were prepared in advance by study personnel, refrigerated, and distributed to study participants on a weekly basis. Participants were provided a daily 32-ounce beverage container for beverage consumption and instructed to clean the container nightly. Participants were asked to keep a log of completion of beverage on a daily basis and instructions regarding intake of other beverages were provided.
- Mediterranean Lemonade: All participants were advised to consume all of the beverage assigned (Mediterranean lemonade) on a daily basis (rather than save up and consume large amounts on fewer days). The beverages were prepared in advance by study personnel, refrigerated, and distributed to study participants on a weekly basis. Participants were provided a daily 32-ounce beverage container for beverage consumption and instructed to clean the container nightly. Participants were asked to keep a log of completion of beverage on a daily basis and instructions regarding intake of other beverages were provided.
- Green Tea: All participants were advised to consume all of the beverage assigned (green tea) on a daily basis (rather than save up and consume large amounts on fewer days). The beverages were prepared in advance by study personnel, refrigerated, and distributed to study participants on a weekly basis. Participants were provided a daily 32-ounce beverage container for beverage consumption and instructed to clean the container nightly. Participants were asked to keep a log of completion of beverage on a daily basis and instructions regarding intake of other beverages were provided.
- Total: Total of all reporting groups
Arm/Group | Flavored Water | Mediterranean Lemonade | Green Tea | Total
Number analyzed (Participants) | 10 | 21 | 19 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (7.1) | 44.5 (9.5) | 48.1 (10.9) | 44.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 15 | 39
  Male | 2 | 5 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mexican | 4 | 11 | 15 | 30
  Mexican-American | 4 | 6 | 3 | 13
  South/Central American | 2 | 1 | 0 | 3
  Other Spanish, Hispanic, Latino | 0 | 2 | 0 | 2
  Missing | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 21 | 19 | 50
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 182.7 (31.6) | 190.5 (45.3) | 200.1 (32.8) | 192.6 (38.2)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dl] | 89.8 (9.8) | 93.0 (12.3) | 93.7 (12.3) | 92.6 (11.7)
Hemoglobin A1C [Mean (Standard Deviation); unit: % of Hemoglobin A1C] | 5.37 (0.28) | 5.52 (0.31) | 5.46 (0.39) | 5.47 (0.34)
Body Weight [Mean (Standard Deviation); unit: kg] | 99.1 (27.9) | 97 (17.7) | 89.9 (15.1) | 94.7 (19.2)

OUTCOME MEASURES:

1. Primary Outcome: Study Recruitment: Interest in Participation
Description: The number of Hispanic adults who contact the researchers and express interest in participation.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Interest in Participation.: The number of Hispanic adults who contact the researchers and express interest in participation.
Arm/Group | Interest in Participation.
Number analyzed (Participants) | 279
Participants | 279

2. Primary Outcome: Study Recruitment: Screened for Eligibility
Description: The number of Hispanic adults screened for eligibility
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Study Recruitment: Screened for Eligibility: The number of Hispanic adults screened for eligibility
Arm/Group | Study Recruitment: Screened for Eligibility
Number analyzed (Participants) | 279
Participants | 236

3. Primary Outcome: Study Recruitment: Eligibility
Description: The number of Hispanic adults eligible for study inclusion.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Study Recruitment: Eligibility: The number of Hispanic adults eligible for study inclusion.
Arm/Group | Study Recruitment: Eligibility
Number analyzed (Participants) | 236
Participants | 104

4. Primary Outcome: Study Recruitment: Ineligibility
Description: The number of Hispanic adults ineligible for study inclusion.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Study Recruitment: Ineligibility: The number of Hispanic adults ineligible for study inclusion.
Arm/Group | Study Recruitment: Ineligibility
Number analyzed (Participants) | 236
Participants | 132

5. Primary Outcome: Enrollment
Description: The number of Hispanic adults enrolled in the study.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Enrollment: The number of Hispanic adults enrolled in the study.
Arm/Group | Enrollment
Number analyzed (Participants) | 104
Participants | 52

6. Primary Outcome: Retention
Description: Retention will be measured as the number of participants who remain in the study at 6 weeks.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Groups:
- Retention: Retention will be measured as the number of participants who remain in the study at 6 weeks.
Arm/Group | Retention
Number analyzed (Participants) | 50
Participants | 44

7. Primary Outcome: Treatment Satisfaction
Description: Participants will be asked to rate their overall satisfaction (1- low; 4-high) with the intervention for changing dietary patterns at Week 6 and if they would recommend the program to others.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment Satisfaction Flavored Water; Treatment Satisfaction Mediterranean Lemonade; Treatment Satisfaction Green Tea: Participants will be asked to rate their overall satisfaction with the intervention for changing dietary patterns at Week 6 and if they would recommend the program to others.
Arm/Group | Treatment Satisfaction Flavored Water | Treatment Satisfaction Mediterranean Lemonade | Treatment Satisfaction Green Tea
Number analyzed (Participants) | 10 | 21 | 19
units on a scale | 3.3 (1.1) | 3.4 (0.9) | 3.3 (1.0)

8. Secondary Outcome: Change in Total Cholesterol (Baseline and Week 6)
Description: Fasting blood samples (venipuncture) will be collected for the purpose of examining changes in total cholesterol.
Time Frame: Baseline and Week 6
Measure: Mean (95% Confidence Interval); unit: mg/dl
Groups:
- Change in Total Cholesterol Flavored Water; Change in Total Cholesterol Mediterranean Lemonade; Change in Total Cholesterol Green Tea: Fasting blood samples (venipuncture) were collected for the purpose of examining changes in total cholesterol.
Arm/Group | Change in Total Cholesterol Flavored Water | Change in Total Cholesterol Mediterranean Lemonade | Change in Total Cholesterol Green Tea
Number analyzed (Participants) | 10 | 21 | 19
mg/dl | -13.2 [-30.2 to 3.8] | -1.67 [-14.2 to 10.9] | -3.9 [-17.2 to 9.4]

9. Secondary Outcome: Change in Fasting Glucose (Baseline and Week 6)
Description: Fasting blood samples (venipuncture) will be collected for the purpose of examining changes in glucose.
Time Frame: Baseline and Week 6
Measure: Mean (95% Confidence Interval); unit: mg/dl
Groups:
- Change in Fasting Glucose Flavored Water; Change in Fasting Glucose Mediterranean Lemonade; Change in Fasting Glucose Green Tea: Fasting blood samples (venipuncture) were collected for the purpose of examining changes in glucose.
Arm/Group | Change in Fasting Glucose Flavored Water | Change in Fasting Glucose Mediterranean Lemonade | Change in Fasting Glucose Green Tea
Number analyzed (Participants) | 10 | 21 | 19
mg/dl | -1.40 [-5.0 to 2.2] | 5.2 [2.6 to 7.9] | 3.3 [0.58 to 6.4]

10. Secondary Outcome: Change in Hemoglobin A1C (Baseline and Week 6)
Description: Fasting blood samples (venipuncture) were collected for the purpose of examining changes in hemoglobin A1C.
Time Frame: Baseline and Week 6
Measure: Mean (95% Confidence Interval); unit: % of Hemoglobin A1C
Groups:
- Change in Hemoglobin A1C Flavored Water; Change in Hemoglobin A1c Mediterranean Lemonade; Change in Hemoglobin A1c Green Tea: Fasting blood samples (venipuncture) were collected for the purpose of examining changes in hemoglobin A1C.
Arm/Group | Change in Hemoglobin A1C Flavored Water | Change in Hemoglobin A1c Mediterranean Lemonade | Change in Hemoglobin A1c Green Tea
Number analyzed (Participants) | 10 | 21 | 19
% of Hemoglobin A1C | -0.02 [-0.14 to 0.1] | 0.05 [-0.04 to 0.14] | 0.04 [-0.06 to 0.14]

11. Secondary Outcome: Change in Body Weight (Baseline and Week 6)
Description: Body weight was measured on a digital scale to assess change in body weight over the intervention period.
Time Frame: Baseline and Week 6
Measure: Mean (95% Confidence Interval); unit: kg
Groups:
- Change in Body Weight Flavored Water; Change in Body Weight Mediterranean Lemonade; Change in Body Weight Green Tea: Body weight was measured on a digital scale to assess change in body weight over the intervention period.
Arm/Group | Change in Body Weight Flavored Water | Change in Body Weight Mediterranean Lemonade | Change in Body Weight Green Tea
Number analyzed (Participants) | 10 | 21 | 19
kg | -1.8 [-2.9 to -0.55] | -0.12 [-1.0 to 0.8] | -0.36 [-1.6 to 1.8]

ADVERSE EVENTS:
Time Frame: 1 year (August 2016-August 2017)
Arm/Group | Mediterranean Lemonade Consumption | Green Tea Consumption | Flavored Water Consumption
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/10
Other Adverse Events (participants affected / at risk) | 2/21 | 0/19 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mediterranean Lemonade Consumption (N=21) | Green Tea Consumption (N=19) | Flavored Water Consumption (N=10)
Gastrointestinal Distress (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was short in duration. It is possible that this was not an adequate amount of time to observe changes in our primary outcomes. In addition, the small sample size may have reduced effect size, thus hindering our capacity to detect changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT02911753/Prot_SAP_000.pdf